CLINICAL TRIAL: NCT03996447
Title: Efficacy and Safety of Gadopiclenol for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)
Acronym: PICTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GDX-44-010
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2023-11

CONDITIONS: CNS Lesion; Blood Brain Barrier Defect
MeSH Terms: interventions — gadopiclenol; gadobutrol; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- gadopiclenol-enhanced MRI then gadobutrol-enhanced MRI (Other): cross-over design. each patient will receive gadopiclenol for the first MRI and gadobutrol for the second MRI
  Interventions: Drug: gadopiclenol; Drug: Gadobutrol 1Mmol/mL Solution for Injection Vial
- gadobutrol-enhanced MRI then gadopiclenol-enhanced MRI (Other): cross-over design. each patient will receive gadobutrol for the first MRI and gadopiclenol for the second MRI
  Interventions: Drug: gadopiclenol; Drug: Gadobutrol 1Mmol/mL Solution for Injection Vial

INTERVENTIONS:
Drug: gadopiclenol — single intravenous (IV) bolus injection at a rate of 2ml/second
Drug: Gadobutrol 1Mmol/mL Solution for Injection Vial — single intravenous (IV) bolus injection at a rate of 2ml/second

SUMMARY:
This trial aimed to evaluate the Efficacy and Safety of gadopiclenol for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)

DETAILED DESCRIPTION:
The purpose of this trial was to evaluate a new gadolinium-based contrast agent (GBCA) gadopiclenol injection for Central Nervous System (CNS) lesion detection and visualization by conventional steady-state CNS imaging.

This is a multi-center, international, prospective, double-blind, randomized, controlled, cross-over with comparator trial in male and female patients presenting with known or highly suspected CNS lesion(s) with focal areas of disrupted Blood Brain Barrier (BBB) (e.g., primary and secondary tumors) who are scheduled to undergo a routine contrast-enhanced Magnetic Resonance Imaging (MRI) of the CNS.

This trial was conducted in 33 centers worldwide.

During the course of the trial, two MRIs were obtained from each patient: one unenhanced and gadopiclenol-enhanced MRI; and one unenhanced and gadobutrol-enhanced MRI. MRI evaluations were performed by on-site investigators and three independent off-site blinded readers.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with known or highly suspected CNS lesion(s) with focal areas of disrupted Blood Brain Barrier (BBB) (e.g., primary and secondary tumors) based on results of a previous imaging procedure such as Computed Tomography (CT) or MRI, which should have been performed within 12 months prior to ICF signature.

Exclusion Criteria:

* Patient presenting with acute or chronic renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m² assessed within 1 day prior to each contrast agent injection
* Patient presenting extra cranial lesions and/or extra-dural lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorie Loevner, MD, Principal Investigator — University of Pennsylvania
Locations (33):
- United States (8):
  - ASCLEPES Research Centers, Panorama City, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwest Neurology, Ltd., Rolling Meadows, Illinois
  - University of Missouri Hospital and Clinic, Columbia, Missouri
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - South Carolina Clinical & Translational Research (SCTR) Institute, Charleston, South Carolina
  - University Of Washington - Medical Center, Seattle, Washington
- Belgium (2):
  - ZNA Middelheim, Antwerp
  - UZ Brussel - Campus Jette, Brussels
- France (4):
  - CHRU - Hôpital Roger Salengro - Neurologie, Lille
  - Centre Hospitalier Sainte-Anne, Paris
  - CHU La Miletrie, Poitiers
  - CHRU Strasbourg Hôpital de Hautepierre, Strasbourg
- Uniklinik Mannheim, Mannheim, Germany
- Hungary (5):
  - Semmelweis Egyetem - Neurology, Budapest
  - Orszagos Klinikai Idegtudomanyi Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont - Idegsebeszeti Klinika, Pécs
  - Szegedi Tudomanyegyetem AOK, Szeged
- Italy (4):
  - ASL 1 Abruzzo Avezzano-Sulmona-L'Aquila, Ospedale Regionale San Salvatore, L’Aquila
  - Fondazione I.R.C.C.S. C.Mondino, Pavia
  - Istituto Neurologico Mediterraneo-Neuromed, I.R.C.C.S., Pozzilli
  - Azienda Sanitaria Universitaria Integrata di Trieste-PO Cattinara, Trieste
- Mexico (2):
  - Axis Heilsa S. de R.L. de C.V. (Althian), Monterrey
  - Clinical Research Institute S.C, Tlalnepantla
- Uniwersyteckie Centrum Kliniczne w Gdańsku, Zakład Radiologii, Gdansk, Poland
- South Korea (2):
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital del Mar, Barcelona
  - M.D. Anderson Cancer Center Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Loevner LA, Kolumban B, Hutoczki G, Dziadziuszko K, Bereczki D, Bago A, Pichiecchio A. Efficacy and Safety of Gadopiclenol for Contrast-Enhanced MRI of the Central Nervous System: The PICTURE Randomized Clinical Trial. Invest Radiol. 2023 May 1;58(5):307-313. doi: 10.1097/RLI.0000000000000944. Epub 2022 Dec 19. PMID 36729404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 260 screened patients, 4 were screen failed. A total of 256 patients were randomized (128 in each arm), of whom 6 discontinued the trial before receiving the first contrast agent. Then 250 patients (125 in each arm) received the first contrast agent and underwent the first MRI (First MRI Period). After a washout period of 2-14 days (Washout Period), 242 patients (120 in the Arm 1 and 122 in the Arm 2) received the second contrast agent and underwent the second MRI (Second MRI Period).
Groups:
- Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadopiclenol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadobutrol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained : unenhanced and gadopiclenol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadobutrol-enhanced MR images obtained in the second MRI Examination Period.
  Gadopiclenol: single intravenous (IV) bolus injection at a rate of 2ml/second
  Gadobutrol 1Mmol/mL Solution for Injection Vial: single intravenous (IV) bolus injection at a rate of 2ml/second
- Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI: Cross-over study design
  For each patient in this Arm, he (she) performed the first contrast-enhanced MRI with gadobutrol as contrast agent (First MRI Period). After a washout period of 2-14 days (Washout Period), the patient performed the second contrast-enhanced MRI with gadopiclenol as contrast agent (Second MRI Period).
  For each patient, two sets of MR images per MRI examination were obtained : unenhanced and gadobutrol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadopiclenol-enhanced MR images obtained in the second MRI Examination Period.
  Gadobutrol 1Mmol/mL Solution for Injection Vial: single intravenous (IV) bolus injection at a rate of 2ml/second
  Gadopiclenol: single intravenous (IV) bolus injection at a rate of 2ml/second
Period: First MRI Examination
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 128 (A total of 256 patients were randomized before first MRI examination: 128 randomized into Arm 1, for whom gadopiclenol-enhanced MRI had to be performed as First MRI examination, and gadobutrol-enhanced MRI to be performed as Second MRI examination.) | 128 (A total of 256 patients were randomized before first MRI examination: 128 randomized into Arm 2, for whom gadobutrol-enhanced MRI had to be performed as the First MRI examination and gadopiclenol-enhanced MRI to be performed as the Second MRI examination.)
Completed | 125 (Among the 128 randomized patients in this arm, 3 patients discontinued the trial before receiving the first contrast agent. Therefore, a total of 125 patients of Arm 1 performed the first MRI examination with gadopiclenol as contrast agent.) | 125 (Among the 128 randomized patients in this arm, 3 patients discontinued the trial before receiving the first contrast agent. Therefore, a total of 125 patients of Arm 2 performed the first MRI examination with gadobutrol as contrast agent.)
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 0 | 1
Period: Washout
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 125 | 125
Completed | 120 (Among the 125 patients in this arm (Arm 1) who performed the MRI with gadopiclenol as contrast agent in the First MRI examination Period, 5 patients discontinued the trial before receiving contrast agent (gadobutrol) for the second MRI.) | 122 (Among the 125 patients in this arm (Arm 2) who performed the MRI with gadobutrol as contrast agent in the First MRI examination Period, 3 patients discontinued the trial before receiving contrast agent (gadopiclenol) for the second MRI.)
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Follow-up unavailable due to COVID-19 pandemic | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other reason | 1 | 1
Period: Second MRI Examination
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI
Started | 120 | 122
Completed | 120 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was based on participants. For the primary analysis to demonstrate the superiority of gadopiclenol-enhanced MRI compared to unenhanced MRI, the analysis population was patients who had both Pre (unenhanced) and Paired (combined unenhanced and contrast-enhanced) images with gadopiclenol assessable for primary criteria for at least one matching lesion for at least one off-site reader: 119 patients of Arm 1 who performed first MRI and 120 patients of Arm 2 who performed second MRI.
Groups:
- Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI: Cross-over study design
  For Arm 1, the patient performed the first contrast-enhanced MRI with gadopiclenol as contrast agent. After a washout period of 2-14 days, the patient performed the second contrast-enhanced MRI with gadobutrol as contrast agent.
  For each patient, two sets of MR images per MRI examination were obtained : unenhanced and gadopiclenol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadobutrol-enhanced MR Images obtained in the Second MRI Examination Period .
- Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI: Cross-over study design
  For Arm 2, the patient performed the first contrast-enhanced MRI with gadobutrol as contrast agent. After a washout period of 2-14 days, the patient performed the second contrast-enhanced MRI with gadopiclenol as contrast agent.
  For each patient, two sets of MR images per MRI examination were obtained : unenhanced and gadobutrol-enhanced MR images obtained in the First MRI Examination Period, unenhanced and gadopiclenol-enhanced MR images obtained in the Second MRI Examination Period.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Gadopiclenol-enhanced MRI for First MRI and Gadobutrol-enhanced MRI for Second MRI | Arm 2: Gadobutrol-enhanced MRI for First MRI and Gadopiclenol-enhanced MRI for Second MRI | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.4) | 56.1 (14.2) | 57.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 63 | 124
  Male | 58 | 57 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 17
  Not Hispanic or Latino | 113 | 109 | 222
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 11 | 16
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 101 | 98 | 199
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 7 | 5 | 12
  Belgium | 2 | 0 | 2
  Hungary | 57 | 43 | 100
  United States | 17 | 24 | 41
  Taiwan | 2 | 2 | 4
  Poland | 11 | 16 | 27
  Italy | 10 | 12 | 22
  Mexico | 5 | 11 | 16
  France | 2 | 4 | 6
  Germany | 1 | 2 | 3
  Spain | 5 | 1 | 6
Weight [Mean (Standard Deviation); unit: Kg] | 77.9 (19.5) | 78.4 (20.8) | 78.1 (20.1)

OUTCOME MEASURES:

1. Primary Outcome: Lesion Visualization Comparing Gadopiclenol-enhanced MRI to Unenhanced MRI
Description: The lesion visualization (per patient) was based on 3 co-primary criteria on marching lesions: border delineation, internal morphology and degree of contrast enhancement, assessed on the images acquired during the MRI performed with gadopiclenol by 3 independent readers. The independent blinded reader recorded each of the 3 co-primary criteria for up to 3 most representative lesions, using a 4-point scale (1 = poor [internal morphology] or none [border delineation, contrast enhancement], 2 = moderate, 3 = good, 4 = excellent). The mean of scores for each patient and for each co-criterion was calculated as follows: Mean of scores = score of lesion 1 + score of lesion 2 (if any) + score of lesion 3 (if any) divided by the number of lesions, ranged from 1 to 4. The difference in mean scores on matching lesions between Paired [unenhanced and contrast-enhanced] images and Pre-contrast [unenhanced] images was calculated for each of the 3 co-primary criteria and for each reader.
Time Frame: At first MRI examination (gadopiclenol-enhanced MRI) for patients of Arm 1. At second MRI examination (gadopiclenol-enhanced MRI) for patients of Arm 2, performed 2-14 days after gadobutrol-enhanced MRI.
Population: Full Analysis Set (FAS) included a total of 239 patients who had both Pre and Paired images with gadopiclenol assessable for primary criteria for at least one matching lesion for at least one off-site reader: 119 patients in the Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 120 patients in the Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI. The analysis was based on participants (per patient).
Measure: Least Squares Mean (Standard Error); unit: mean of a score (on a scale) per patient
Groups:
- Patients With Gadopiclenol Paired Images: The analysis included 239 patients on marching lesions who had both gadopiclenol Paired images and gadopiclonol Pre images:
  119 patients of Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 120 patients of Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI.
  The analysis was based on participants (at patient level).
  Therefore, the 239 patients with gadopiclenol Paired images are the same patients with gadopiclenol Pre images.
- Patients With Gadopiclenol Pre Images: The analysis included 239 patients on marching lesions who had both gadopiclenol Paired images and gadopiclonol Pre images:
  119 patients of Arm 1 for whom gadopiclenol-enhanced MRI was performed as first MRI, and 120 patients of Arm 2 for whom gadopiclenol-enhanced MRI was performed as second MRI.
  The analysis was based on participants (at patient level).
  Therefore, the 239 patients with gadopicleno Pre images are the same patients with gadopiclenol Paired images.
Arm/Group | Patients With Gadopiclenol Paired Images | Patients With Gadopiclenol Pre Images
Number analyzed (Participants) | 239 | 239
mean of a score (on a scale) per patient
  Border delineation - Reader 1 | 3.90 (0.02) | 2.08 (0.02)
  Border delineation - Reader 2 | 3.64 (0.04) | 1.74 (1.90)
  Border delineation - Reader 3 | 3.97 (0.03) | 2.61 (0.03)
  Internal morphology - Reader 1 | 3.92 (0.03) | 1.66 (0.03)
  Internal morphology - Reader 2 | 3.65 (0.03) | 1.88 (0.03)
  Internal morphology - Reader 3 | 3.97 (0.04) | 2.01 (0.04)
  Contrast enhancement - Reader 1 | 3.77 (0.03) | 1.00 (0.03)
  Contrast enhancement - Reader 2 | 3.58 (0.03) | 1.00 (0.03)
  Contrast enhancement - Reader 3 | 3.90 (0.02) | 1.00 (0.02)
Statistical Analysis 1: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 1. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error set at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously and for at least 2 out of 3 readers; Test type: Superiority; p < .0001, t-test, 2 sided — To demonstrate the superiority, a statistically significant (one-sided p-value ≤0.025) positive difference in mean scores in border delineation, internal morphology and degree of contrast enhancement of lesions had to be met for 2 out of 3 readers; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [1.76 to 1.88], Standard Error of Mean 0.03
Statistical Analysis 2: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 2. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [1.81 to 2.00], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Border delineation; Reader 3. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.36, 95% CI 2-sided [1.29 to 1.44], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 1. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [2.20 to 2.33], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 2. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [1.69 to 1.85], Standard Error of Mean 0.04
Statistical Analysis 6: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Internal morphology; Reader 3. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [1.85 to 2.06], Standard Error of Mean 0.05
Statistical Analysis 7: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement; Reader 1. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.77, 95% CI 2-sided [2.69 to 2.85], Standard Error of Mean 0.04
Statistical Analysis 8: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement - Reader 2. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.58, 95% CI 2-sided [2.49 to 2.67], Standard Error of Mean 0.05
Statistical Analysis 9: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadopiclenol Pre Images; Criterion: Contrast enhancement; Reader 3. The null hypothesis was that the difference in mean scores between Paired images and Pre-contrast images for each of the 3 co-primary criteria was equal to 0. The Null hypothesis was rejected if the difference was significantly different from zero with a type 1 error at 0.025. To conclude the superiority of gadopiclenol-enhanced MRI, the null hypothesis had to be rejected for all co-criteria simultaneously; Test type: Superiority; p < .0001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.90, 95% CI 2-sided [2.84 to 2.95], Standard Error of Mean 0.03

2. Secondary Outcome: Lesion Visualization Comparing Gadopiclenol-enhanced MRI to Gadobutrol-enhanced MRI
Description: The lesion visualization (per patient) was based on 3 co-primary criteria: border delineation, internal morphology and degree of contrast enhancement, assessed on the images performed with gadopiclenol and images performed with gadobutrol by 3 independent readers. The independent blinded reader recorded each of the 3 co-primary criteria for up to 3 most representative lesions, using a 4-point scale (1 = poor [internal morphology] or none [border delineation, contrast enhancement], 2 = moderate, 3 = good, 4 = excellent). The mean of scores for each patient and for each of the 3 lesion visualization co-criteria was calculated as follows: Mean of scores = score of lesion 1 + score of lesion 2 (if any) + score of lesion 3 (if any) divided by the number of lesions, ranged from 1 to 4. The difference in mean scores on matching lesions between gadopiclenol scores mean and gadobutrol scores mean was calculated for each of the 3 co-primary criteria and for each reader.
Time Frame: At each of two MRI examinations with an interval of 2-14 days between 2 MRI examinations
Population: Per-Protocol Set (PPS) analysis population including a total of 236 patients (117 patients of Arm 1 and 119 patients of Arm 2) with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader. The analysis was based on participants (per patient).
Measure: Least Squares Mean (Standard Error); unit: mean of a score (on a scale) per patient
Groups:
- Patients With Gadopiclenol Paired Images: Analysis included 236 patients (117 patients in the Arm 1 and 119 patients in the Arm 2) with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader:
  The analysis was based on participants (per patient).
  The 236 patients with gadopiclenol Paired images are the same patients with gadobutrol Paired images.
- Patients With Gadobutrol Paired Images: Analysis included 236 patients (117 patients in the Arm 1 and 119 patients in the Arm 2) with no major protocol deviation who have Paired (combined unenhanced and contrast-enhanced) images for both gadopiclenol and gadobutrol assessable for this secondary outcome mesure for at least one matching lesion for at least one off-site reader:
  The analysis was based on participants (per patient).
  The 236 patients with gadobutrol Paired images are the same patients with gadopiclenol Paired images.
Arm/Group | Patients With Gadopiclenol Paired Images | Patients With Gadobutrol Paired Images
Number analyzed (Participants) | 236 | 236
mean of a score (on a scale) per patient
  Border delineation - Reader 1 | 3.91 (0.02) | 3.93 (0.02)
  Border delineation - Reader 2 | 3.64 (0.04) | 3.60 (0.04)
  Border delineation - Reader 3 | 3.97 (0.01) | 3.95 (0.01)
  Internal morphology - Reader 1 | 3.93 (0.02) | 3.93 (0.02)
  Internal morphology - Reader 2 | 3.64 (0.04) | 3.62 (0.04)
  Internal morphology - Reader 3 | 3.97 (0.02) | 3.92 (0.02)
  Contrast enhancement - Reader 1 | 3.78 (0.04) | 3.77 (0.04)
  Contrast enhancement - Reader 2 | 3.57 (0.04) | 3.52 (0.04)
  Contrast enhancement - Reader 3 | 3.89 (0.03) | 3.81 (0.03)
Statistical Analysis 1: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 1. The null hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 primary criteria was equal to the non inferiority margin (-0.35). The alternative hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 co-primary criteria was greater than the non inferiority margin; Test type: Non-Inferiority — Non-inferiority between gadopiclenol and gadobutrol was concluded if the lower bound of this confidence interval was above the non-inferiority margin set to 0.35 for at least 2 out of 3 blinded readers and for the 3 co-primary criteria simultaneously; p < 0.0001, t-test, 2 sided — The Null hypothesis was rejected if the 2-sided 95% Confidence Interval (CI) for the difference [gadopiclenol scores mean - gadobutrol scores mean] had its lower limit above -0.35; The Student's t-based 95% CIs of the difference between gadopiclenol and gadobutrol were constructed for each of 3 co-primary criteria; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.02], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 2. The null hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 primary criteria was equal to the non inferiority margin (-0.35). The alternative hypothesis was that the difference in mean scores between gadopiclenol and gadobutrol for each of the 3 co-primary criteria was greater than the non inferiority margin; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.04 to 0.11], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Border delineation; Reader 3; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.05], Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 1; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.04 to 0.03], Standard Error of Mean 0.02
Statistical Analysis 5: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 2; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.05 to 0.09], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Internal morphology; Reader 3; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.01 to 0.08], Standard Error of Mean 0.02
Statistical Analysis 7: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 1; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.04 to 0.07], Standard Error of Mean 0.03
Statistical Analysis 8: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 2; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.03 to 0.12], Standard Error of Mean 0.04
Statistical Analysis 9: Comparison: Patients With Gadopiclenol Paired Images vs Patients With Gadobutrol Paired Images; Criterion: Contrast enhancement; Reader 3; Test type: Non-Inferiority — Non-inferiority margin : -0.35; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [0.03 to 0.15], Standard Error of Mean 0.03

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from informed consent signature up to one day after the second MRI (i.e., minimum of 4 days and a maximum of 23 days)
Groups:
- Gadopiclenol: AEs reported after MRI with gadopiclenol
- Gadobutrol: AEs reported after MRI with gadobutrol
Arm/Group | Gadopiclenol | Gadobutrol
All-Cause Mortality (participants affected / at risk) | 0/247 | 1/245
Serious Adverse Events (participants affected / at risk) | 0/247 | 1/245
Other Adverse Events (participants affected / at risk) | 36/247 | 42/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadopiclenol (N=247) | Gadobutrol (N=245)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1) — Not related to contrast-agent
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadopiclenol (N=247) | Gadobutrol (N=245)
Injection site pain (General disorders) | 5 (5) | 5 (5)
Injection site bruising (General disorders) | 3 (3) | 3 (3)
Injection site erythema (General disorders) | 1 (1) | 3 (3)
Injection site coldness (General disorders) | 2 (2) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 2 (2)
Injection site haematoma (General disorders) | 1 (1) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (2)
Injection site paraesthesia (General disorders) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 2 (5)
Asthenia (General disorders) | 0 (0) | 1 (1)
Drug ineffective (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Partial seizures (Nervous system disorders) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 5 (5)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT03996447/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03996447/SAP_001.pdf